CLINICAL TRIAL: NCT05549973
Title: Single-center, Open-label, Single-arm Exploratory Clinical Trial of Anlotinib Monotherapy and Combination Therapy in Relapsed / Refractory MM Previously Treated With Immunomodulator and Protease Inhibitor Regimens
Brief Title: Anlotinib Hydrochloride Capsule Monotherapy and Combination Therapy Relapsed and Refractory Multiple Myeloma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Principal Investigator, Gang An, Deputy Chief Physician, Institute of Hematology & Blood Diseases Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: An-MM-001
Record Dates: First submitted 2022-09-07; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib Hydrochloride Capsule (Experimental): Anlotinib Hydrochloride Capsule, 21 days as a treatment cycle.
  Interventions: Drug: Anlotinib Hydrochloride Capsule

INTERVENTIONS:
Drug: Anlotinib Hydrochloride Capsule — Anlotinib hydrochloride is a muti-target tyrosine kinase inhibitor.
  Other Names: dexamethasone

SUMMARY:
This is a Single-center, Open-label, Single-arm Exploratory Clinical Study to evaluate the safety and efficacy of Anlotinib Hydrochloride Capsule Monotherapy and Combination Therapy in relapsed or refractory multiple myeloma patient.

DETAILED DESCRIPTION:
This study is an exploratory study, which is divided into two parts. The first part uses BOIN design to explore the phase II recommended dose and safety of anlotinib monotherapy or combination regimen. The second part explored the efficacy and safety of anlotinib in the treatment of RRMM with phase II recommended dose monotherapy and combination regimen. Set up two treatment options, in which A program for monotherapy : Anlotinib monotherapy + dexamethasone ; regimen B is a combination therapy regimen : anlotinib combined with pomalidomide or dalattoumab + dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

1. known and volunteered to sign the Informed Consent;
2. Age≥ 18 years
3. Patients must have previously received a regimen containing immunomodulators and protease inhibitors, and the end-line treatment regimen is refractory or intolerant ( patients recorded as intolerant must discuss and obtain permission from the sponsor 's medical inspector before entering the screening ). Refractory includes primary refractory ( patients did not achieve minimal remission MR or disease progression during treatment ) or secondary refractory ( patients developed disease progression within 60 days after treatment ).
4. Non-hematological toxicity associated with previous treatment occurring prior to the first use of the drug must be reduced to ≤ grade 2, except for peripheral neuropathy, which is specified in article 17 of the exclusion criteria.
5. Liver function met the following criteria : total bilirubin < 2 × upper limit of normal range ( ULN ) ( for patients with Gilbert syndrome, total bilirubin < 3 × ULN ), AST < 2.5 × ULN and ALT < 2.5 × ULN.
6. Renal function meets the following criteria : creatinine clearance ≥ 20 mL / min ( Cockroft-Gault formula ).
7. The ECOG performance status score is 0, 1 or 2.
8. With measurable multiple myeloma, at least one of the following needs to be met :

   1. Serum M protein ( SPEP ) ≥ 5 g / L.
   2. 24 hour urinary M protein excretion rate ≥ 0.2g ( 200mg ).
   3. Serum free light chain ( sFLC ) ≥ 100 mg / L and abnormal free light chain ratio.
9. Blood routine examination met the following criteria ( platelet transfusion was not received within 1 week before the first study, and red blood cell transfusion was not received within 2 weeks before the first study ) :

   1. Hemoglobin level ≥ 80g / L.
   2. Absolute neutrophil count ( ANC ) ≥ 1000 / mm3 ( 1.0x109 / L ).
   3. If the proportion of plasma cells in bone marrow < 50 %, platelet count ≥ 75,000 / mm3 ( 75x109 / L ) ; such as bone marrow plasma cell ratio ≥ 50 %, platelet count ≥ 50,000 / mm3 ( 50x109 / L ).

   10.10.Possible pregnant women must meet the following two conditions :

   a. Agrees to use both contraceptive methods approved by the research physician or complete abstinence during the use of the research drug and within three months after the last administration of the research drug from the date of signing the informed consent.

   i. Abstinence : Acceptable when this method is consistent with the preferred and daily lifestyle of the subject. Periodic abstinence ( such as according to the calendar, ovulation, symptoms of body temperature, after ovulation method ) is not accepted.

   ii. acceptable contraceptive methods include : oral contraceptives, injectable contraceptives or implantable hormonal contraceptives ; intrauterine device ; barrier contraceptive tools with spermicide ; or the partner received sterilization, combined with the use of at least one barrier contraceptive.

   b. screening serum pregnancy test results were negative. Note : Fertility refers to all women who have begun their menstrual period, are not in the post-menopausal period and have not undergone surgical sterilization ( e.g. hysterectomy, bilateral tubal ligation, bilateral ovariectomy ). Postmenopause refers to amenorrhea for more than 12 consecutive months for non-specific reasons. Women who are using mechanical contraceptive methods such as oral contraceptives or intrauterine devices should be considered to have fertility.

11. Male subjects ( including those who have undergone vasectomy ) must consent to the use of condoms in their sexual life with women of childbearing age and, from the date of signing the informed consent form, have no plans to conceive a woman during the use of the study drug and within three months after the last administration of the study drug.

Exclusion Criteria:

1. Asymptomatic ( smoking ) multiple myeloma.
2. Plasma cell leukemia.
3. Clarify the combined amyloidosis.
4. Multiple myeloma with central nervous system ( CNS ) invasion.
5. Pregnancy or lactation.
6. First study before medication A. Receiving chemotherapy within 1 week. b. received radiotherapy or immunotherapy within 4 weeks. c. Radioimmunotherapy within 6 weeks.
7. Transplant rejection ( after allogeneic stem cell transplantation ).
8. Life expectancy < 4 months.
9. Oversized surgery within 4 weeks before first study medication.
10. Patients with unstable or active cardiovascular diseases, in line with any of the following :

    1. Symptomatic myocardial ischemia ;
    2. Uncontrolled and clinically significant conduction abnormalities ( e.g., exclusion of patients with ventricular arrhythmias controlled by antiarrhythmic drugs ; patients with 1 degree atrioventricular ( AV ) block or asymptomatic left anterior bundle branch block / right bundle branch block ( LAFB / RBBB ) were not excluded.
    3. New York Heart Association ( NYHA ) definition of congestive heart failure ( CHF ) classification ≥ 3 ;
    4. Acute myocardial infarction ( AMI ) occurred within 3 months before the first study.
11. Poorly controlled hypertension ( persistent systolic > 140 mmHg or diastolic > 90 mmHg ).
12. In the first study, there were active infections that were not effectively controlled by drugs within 1 week before treatment.
13. Known HIV positive.
14. A, B, C hepatitis infection active period or known HCV RNA or HBsAg ( HBV surface antigen ) positive.

    Note : Including HBsAg negative but hepatitis B core ( HBc ) antibody positive, and detectable levels of hepatitis B virus deoxyribonucleic acid ( HBV-DNA ) ( HBV-DNA > 500 IU / ml ).
15. In the 5-year period before the first study, there were previous malignant tumors that needed treatment or had evidence of recurrence [ except for skin basal cell carcinoma and the following carcinoma in situ : squamous cell carcinoma, bladder carcinoma in situ, endometrial carcinoma in situ, cervical carcinoma in situ / atypical hyperplasia, incidental histological findings of prostate cancer ( TNM stage T1a or T1b ) or breast carcinoma in situ ].
16. There is dysphagia or active gastrointestinal ( GI ) dysfunction that may affect drug absorption.
17. There were ≥ grade 3 peripheral neuropathy and ≥ grade 2 painful neuropathy within 3 weeks before the first study.
18. Active mental disorders or organic diseases considered by researchers to be unsuitable for inclusion.
19. Participated in clinical trials of other drugs within three weeks or five drug half-lives ( T1 / 2 ) prior to the first study.
20. Before treatment received the following treatment, in line with any of the following :

    1. Platelet transfusion within 1 week before the first study ;
    2. infusion of red blood cells ( RBC ) within 2 weeks before the first study ;
    3. The following blood growth factors were used within 2 weeks prior to the first study : granulocyte colony-stimulating factor ( G-CSF ), granulocyte-macrophage colony-stimulating factor ( GM-CSF ), erythropoietin ( EPO ), megakaryocyte growth factor, and / or platelet-stimulating factor.
21. Intolerance or contraindications to glucocorticoid therapy are known.
22. Anlotinib has been used.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Overall response rate ( ORR ) | From date of randomization until the date of first documented progression,assessed up to 100 months
  partial remission ( PR ) + very good partial remission ( VGPR ) + complete remission ( CR ) + strict complete remission ( sCR ).

SECONDARY OUTCOMES:
6 months, 9 months, 12 months survival rate ( SR ) | 6 months, 9 months, 12 months
  6 months, 9 months, 12 months survival rate
TTP | From date of randomization until the date of death from any cause,assessed up to 100 months
  Duration from treatment initiation to disease progression
PFS | From date of randomization until the date of death from any cause,assessed up to 100 months
  Time from the start of treatment to disease progression or death from any cause
DOR | From date of randomization until the date of death from any cause,assessed up to 100 months
  Duration from first observation of at least partial remission ( PR ) to disease progression or death from disease progression, whichever comes first
CBR | From date of randomization until the date of death from any cause,assessed up to 100 months
  ORR + Minimal Remission ( MR )
Clinical Benefit Rate ( CBR ) + Stable Disease DCR | 12 weeks
  clinical benefit rate ( CBR ) + stable disease ( SD : at least 12 weeks )
OS | From date of randomization until the date of death from any cause,assessed up to 100 months
  Time from initiation of treatment to death from any cause
MRD in CR and sCR patients MRD in CR and sCR patients | through study completion, an average of 1 year
  Minimal residual disease ( MRD ) in patients with CR or sCR
The influence of risk factors stratification based on fluorescence in situ hybridization ( FISH ) on clinical efficacy, including del 13, del 17p13, t ( 4 ; 14 ), t ( 14 ; 16 ), 1q21 amplification | 28 days
  FISH analysis to diagnose and determine MM subtypes
security of medical | From date of randomization until the date of first documented progression,assessed up to 100 months
  Including hematological toxicity and non-hematological toxicity ; neutropenia, thrombocytopenia, anemia and hand-foot skin reaction, hypertension, hypertriglyceridemia, proteinuria, diarrhea, fatigue, hemoptysis, hypothyroidism, hyponatremia, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Gang An, Principal Investigator — chief physician
Locations (1):
- InstituteHBDH, Tianjin, Tianjin Municipality, China